CLINICAL TRIAL: NCT06293287
Title: Enoxaparin for Preventing the Radical Artery Occlusion After the Transradial Access Hepatic Arterial Infusion Chemotherapy: A Multicenter, Randomized Controlled Trial.
Brief Title: Enoxaparin for Preventing the Radical Artery Occlusion After the Transradial Access Hepatic Arterial Infusion Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital (Xiamen), Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DJ-2023-02
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-01

CONDITIONS: Radial Artery Occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The control group will receive an injection of a placebo (0.9% saline solution) of equal volume once daily.
  Interventions: Drug: Placebo
- enoxaparin sodium (Active Comparator): Subjects in the experimental group will be administered subcutaneous enoxaparin sodium injections at a dose of 4000 Axa IU once daily.
  Interventions: Drug: Subcutaneous enoxaparin sodium

INTERVENTIONS:
Drug: Subcutaneous enoxaparin sodium — Subcutaneous enoxaparin sodium injections at a dose of 4000 Axa IU once daily
  Arms: enoxaparin sodium
Drug: Placebo — placebo (0.9% saline solution)
  Arms: placebo

SUMMARY:
The present investigation is designed as a single-blind, randomized, controlled, bicentric trial. The objective is to ascertain whether the subcutaneous administration of enoxaparin sodium for prophylactic anticoagulation during transradial hepatic arterial infusion chemotherapy (HAIC) can diminish the incidence of radial artery occlusion (RAO) post-procedure

DETAILED DESCRIPTION:
Primary liver cancer ranks sixth globally in incidence and fourth in mortality, with over 800,000 new cases annually . Hepatocellular carcinoma (HCC) accounts for over 80% of primary liver cancers. Due to its insidious onset, most patients present with intermediate to advanced stage disease at diagnosis and are ineligible for curative treatments such as surgical resection or liver transplantation. For unresectable liver cancer, a combination of locoregional therapies (e.g., transarterial chemoembolization, hepatic arterial infusion chemotherapy) and systemic treatments (e.g., targeted therapy, immunotherapy) constitute the standard care.

Hepatic Arterial Infusion Chemotherapy (HAIC) delivers high concentrations of chemotherapy agents directly to the tumor via the hepatic artery, leading to more effective tumor cell kill and suppression. Recent advances in HAIC using the FOLFOX regimen (oxaliplatin, fluorouracil) for intermediate and advanced HCC have been made by researchers in China . However, HAIC typically requires long infusion times. Traditional HAIC involves arterial sheath and catheter placement via the femoral artery, necessitating bed rest for 24-48 hours post-operation, reducing patient comfort, and increasing the risk of deep vein thrombosis in the lower limbs due to prolonged immobilization . Recently, the transradial approach for peripheral intervention has gained attention. Transradial HAIC is favored in clinical practice as it does not require postoperative immobilization or carry the risk of causing deep vein thrombosis in the lower limbs.

Radial artery occlusion (RAO) is the most common complication following transradial interventions, often asymptomatic and diagnosed via radial artery ultrasound. The incidence of RAO post-transradial coronary interventions is reported to be between less than 1% to 33% . Preventive measures for RAO typically include: using catheters of the appropriate size (sheath diameter should be less than the radial artery lumen); intraoperative use of unfractionated heparin, short-term postoperative oral anticoagulation; patent hemostasis and shorter compression times . Transradial HAIC is a relatively new practice with limited research. A recent domestic study indicated that the incidence of RAO following transradial FOLFOX-HAIC was as high as 35%, potentially related to prolonged sheath placement and multiple procedures. Retrospective and prospective analyses suggest that the use of low molecular weight heparin during infusion may reduce the incidence of RAO postoperatively . While prophylactic anticoagulation is standard for patients at high risk of venous thromboembolism, it is not typically administered to low-risk patients. Hence, the potential of enoxaparin sodium for prophylactic anticoagulation during transradial HAIC to reduce RAO incidence warrants further investigation.

RAO can preclude the possibility of future transradial interventions, impacting the patient's options for intervention access and treatment strategy. Thus, preventing RAO following transradial HAIC has significant clinical importance. This study aims to explore the efficacy of prophylactic enoxaparin sodium in preventing postoperative RAO through a randomized controlled trial.

Case Number and Grouping Method:

This study plans to recruit 156 subjects and will use a 1:1 randomization to divide them into an experimental group and a control group.

Participant Data Collection and Randomization:

Data will be collected from subjects on radial artery Doppler ultrasound, coagulation function, and complete blood count within one week prior to receiving trans-radial FOLFOX-HAIC. Those who meet the inclusion criteria will be randomized into the experimental group or the control group in a 1:1 ratio. Specifically, each participant will be assigned a unique identification code, and a random number generator will be used for random allocation to the different treatment groups. This process will be computerized, unpredictable, and uncontrollable, ensuring an equal probability of assignment to each group, known as "randomization." The study will be blind to the subjects.

For anticoagulation during trans-radial HAIC chemotherapy, there are no unified clinical guidelines on whether routine prophylactic anticoagulation is necessary. Enoxaparin sodium is a commonly used clinical anticoagulant for the prevention and treatment of thromboembolic disorders, including deep vein thrombosis. Past research has suggested that the use of enoxaparin sodium during HAIC may reduce the incidence of postoperative RAO (Radial Artery Occlusion). After the trans-radial HAIC treatment and catheter removal, subjects in the experimental group will be administered subcutaneous enoxaparin sodium injections at a dose of 4000 Axa IU once daily, while the control group will receive an injection of a placebo (0.9% saline solution) of equal volume once daily. After sheath removal, compression will be applied for two hours before being relieved.

During the treatment with low-molecular-weight heparin, patients will be closely monitored for any signs of bleeding, such as from the skin, mucous membranes, gum bleeding, or black stools. On the first day after the procedure, routine blood counts and coagulation function will be checked. Radial artery Doppler ultrasounds will be performed 24 hours later and again after 21 days to assess for the occurrence of RAO. In case of RAO, anticoagulant therapy will be administered promptly.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent; Age: 18-69 years;
2. Pathologically diagnosed with hepatocellular carcinoma or clinically in accordance with the American Association for the Study of Liver Diseases (AASLD) diagnostic criteria for hepatocellular carcinoma;
3. Clinical stage: BCLC stage B or C, liver function Child-Pugh class A or B$ (≤7 points)$, ECOG $score <2$; suitable for HAIC treatment;
4. Adequate hematological and organ function, i.e., based on laboratory results obtained within 7 days before treatment, such as complete blood count, liver and kidney function, coagulation function, myocardial enzymes, etc., to assess whether the patient is suitable for HAIC treatment;
5. Low-risk patients for VTE (Venous Thromboembolism) according to the Padua scoring system (≤3 points).

Exclusion Criteria:

1. Concomitant primary tumors of other organs or histologically diagnosed tumors inconsistent with hepatocellular carcinoma;
2. Serious diseases of the heart, lungs, kidneys, or other organs;
3. Patients who have received trans-radial interventional surgery within the past 3 months;
4. Patients with thrombocytopenia $and/or $leukopenia due to cirrhosis-related coagulation disorders or splenic hyperfunction are excluded;
5. Preoperative radial artery ultrasound suggests vascular anatomical abnormalities, malformations, etc., unsuitable for trans-radial interventional treatment;
6. Patients with thrombotic diseases who are undergoing anticoagulation therapy;
7. Any unstable conditions or situations that may jeopardize the patient's safety or their compliance with the study;
8. Pregnant and lactating women.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
RAO rate after 24 hours and 21days | Data will be analyzed immediately after the last participant completes the 21-day post-treatment radial artery Doppler ultrasound assessment.
  Radial artery Doppler ultrasounds will be performed 24 hours later and again after 21 days to assess for the occurrence of RAO.

CONTACTS AND LOCATIONS:
Overall Officials: BoHeng Zhang, PHD, Study Chair — Zhongshan Hospital (Xiamen), Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University (Xiamen Branch), Xiamen, Fujian, China